CLINICAL TRIAL: NCT01031355
Title: Open-label, Randomized, Cross-over Study to Investigate the Bioequivalence of Estradiol Valerate (EV) and Levomefolate Calcium After Single Oral Administration of a Tablet Formulation Containing 3 mg EV Without and With 0.451 mg Levomefolate Calcium and a Tablet Formulation Containing 0.451 mg Levomefolate Calcium in 42 Healthy Postmenopausal Women
Brief Title: Bioequivalence Study: 3 mg Estradiol Valerate (EV) With and Without Levomefolate Calcium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13468; 2009-011962-27 (EudraCT Number)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Contraception; Ovulation Inhibition
Keywords: Female Contraception; Contraceptives, Oral
MeSH Terms: interventions — Estradiol; levomefolate calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Estradiol Valerate (EV) / Levomefolate Calcium (BAY98-7078)
- Arm 2 (Active Comparator)
  Interventions: Drug: Estradiol Valerate (EV) (BAY86-4980)
- Arm 3 (Active Comparator)
  Interventions: Drug: Levomefolate Calcium (BAY86-7660)

INTERVENTIONS:
Drug: Estradiol Valerate (EV) / Levomefolate Calcium (BAY98-7078) — Oral, single dose, 3 mg EV + 0.451 mg levomefolate calcium, washout phase between treatments: at least 7 days
  Arms: Arm 1
Drug: Estradiol Valerate (EV) (BAY86-4980) — Oral, single dose, 3 mg EV, washout phase between treatments: at least 7 days
  Arms: Arm 2
Drug: Levomefolate Calcium (BAY86-7660) — Oral, single dose, 0.451 mg levomefolate calcium, washout phase between treatments: at least 7 days
  Arms: Arm 3

SUMMARY:
Investigation of the bioequivalence (BE) of Estradiol Valerate (EV) after administration of one film-coated tablet containing 3 mg Estradiol Valerate and 0.451 mg Levomefolate calcium as compared to one film-coated tablet containing 3 mg Estradiol Valerate Investigation of the bioequivalence of levomefolate calcium after administration of one film-coated tablet containing 3 mg Estradiol Valerate and 0.451 mg Levomefolate calcium as compared to one film-coated tablet containing 0.451 mg levomefolate calcium

ELIGIBILITY:
Inclusion Criteria:

* BMI:>18 <30 kg/m²
* Healthy female volunteers
* Age 45-75 years
* Postmenopausal state

Exclusion Criteria:

* Contraindications for use of combined (Estradiol Valerate/dienogest) contraceptive (e.g.history of venous/arterial thromboembolic disease)
* Regular intake of medication
* Clinically relevant findings (ECG, blood pressure, physical and gynaecological examination, laboratory examination)
* Smoking

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Uncorrected Cmax and AUC(0-tlast) and baseline corrected Cmax and AUC (if possible) for E1, E2, E1S, and L-5- methyl-THF | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Neu-Ulm, Bavaria, Germany